CLINICAL TRIAL: NCT00597493
Title: Phase 2 Study of Sorafenib Plus Protracted Temozolomide in Recurrent Glioblastoma Multiforme
Brief Title: Ph. 2 Sorafenib + Protracted Temozolomide in Recurrent GBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bayer (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000464
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: Recurrent Glioblastoma Multiforme; GBM; Glioblastoma; Sorafenib; Temozolomide; Brain Tumor; Recurrent GBM; Temodar; Gliosarcoma; Glioma; Nexavar
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Gliosarcoma; Glioma | interventions — Sorafenib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib + Temozolomide (Experimental): Subjects receive 400mg of Sorafenib twice daily and 50mg/m^2 of Temozolomide once daily
  Subjects continue to receive treatment until any of the following: progressive disease, unacceptable toxicity, non-compliance with study guidelines, withdrawal of patient consent, intercurrent non-cancer-related illness that prevents continuation of therapy or regular follow-up, general or specific changes in a subject's condition which render the patient unacceptable for treatment in the judgement of the investigator, or study closure
  Interventions: Drug: Sorafenib and Temozolomide

INTERVENTIONS:
Drug: Sorafenib and Temozolomide — Temozolomide (50 mg per meter-squared of body surface area)every day by mouth in combination with sorafenib. Sorafenib will be taken by mouth twice every day. The dose of sorafenib will be 400 mg (2 x 200mg tablets).
  Other Names: Temodar; Nexavar

SUMMARY:
PURPOSE AND OBJECTIVES:

Primary Objective To evaluate the activity of Sorafenib plus protracted, daily temozolomide in patients with recurrent glioblastoma multiforme (GBM) as measured by 6-month PFS.

Secondary Objectives To evaluate the safety and toxicity of combination therapy using Sorafenib plus temozolomide; To determine the pharmacokinetics of Sorafenib when combined with temozolomide in patients on and not on concurrent EIAC medications.

DETAILED DESCRIPTION:
STUDY ACTIVITIES AND POPULATION GROUP:

This is an open-label, non-randomized, single center phase 2 trial. A treatment cycle will consist of 4 weeks of therapy.

Sorafenib will be administered at a set dose of 400 mg (2 x 200 mg tablets) twice daily, without food (at least 1 hour before or 2 hours after eating). Temozolomide will be administered at a set dose of 50 mg/m2 once daily without food (at least 1 hour before or 2 hours after eating).

Thirty-two (32) patients will be enrolled in this single-stage study.

DATA ANALYSIS AND RISK/SAFETY ISSUES:

After 16 patients with recurrent GBM are treated, an interim analysis will be conducted. If 6 or more patients have experienced unacceptable toxicity, accrual of patients in this patient group will be terminated. Otherwise, patient accrual will continue. If 9 or more of the total 32 patients experience unacceptable toxicity, the treatment regimen will be considered to have an unacceptable toxicity profile. The type I and II error rates associated with this testing are 0.053 and 0.053, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of recurrent/progressive GBM. Recurrence will be distinguished from "pseudoprogression" following XRT/Temodar as outlined in inclusion criteria 4.6 (below). Pts with recurrent disease whose diagnostic pathology confirmed glioblastoma multiforme will not need re-biopsy. Pts with prior low-grade glioma or WHO grade III malignant glioma are eligible if histologic assessment demonstrates transformation to GBM.
* Age > 18 years.
* Pts must be presenting in 1st, 2nd or 3rd relapse. Prior therapy must have included external beam radiotherapy.
* Adequate bone marrow, liver and renal function as assessed by following:

  * Hemoglobin > 9.0 g/dl
  * Absolute neutrophil ct (ANC) > 1,500/mm3
  * Platelet ct > 100,000/mm3
  * Total bilirubin < 1.5 x ULN
  * ALT & AST < 2.5 x ULN ( < 5 x ULN for pts with liver involvement)
  * INR < 1.5 or PT/PTT within normal limits (unless on therapeutic anti-coagulation). Pts receiving anti-coagulation treatment with agent such as warfarin or heparin may be allowed to participate. For pts on warfarin, INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by local standard of care, until INR is stable.
  * Creatinine < 1.5 x ULN
* An interval of at least 2 weeks between prior surgical resection (1 week for biopsy)& initiation of study regimen;
* An interval of at least 12 weeks from completion of standard, daily XRT, unless 1 of the following occurs: 1) new area of enhancement on MRI imaging that is outside XRT field; 2) biopsy proven recurrent tumor; 3) radiographic evidence of progressive tumor on 2 consecutive scans at least 4 weeks apart.
* An interval of at least 4 weeks from prior chemotherapy (except nitrosoureas which require 6 weeks) unless there is unequivocal evidence of tumor progression and pts has recovered from all anticipated toxicities from prior therapy.
* Karnofsky performance score > 60%.
* Ability to understand and willingness to sign written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* If sexually active, patients will take contraceptive measures (barrier method of birth control) for duration of treatments and for 3 months following discontinuation of sorafenib & temozolomide.
* Pts who have had prior bevacizumab are eligible however interval of at least 6 weeks must have elapsed since their last dose.

Exclusion Criteria:

* Prior treatment with sorafenib.
* Significant cardiac disease including any of following: a) congestive heart failure > class II NYHA; b) unstable angina (anginal symptoms at rest); c) new onset angina (within last 3 months); d) myocardial infarction within past 6 months; e) cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Known severe hypersensitivity to sorafenib or any of excipients or temozolomide.
* Excessive risk of bleeding as defined by stroke within prior 6 months, history of CNS or intraocular bleed, or septic endocarditis.
* Female pts who are pregnant/breast feeding, or adults of reproductive potential not employing effective method of birth control.
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in study such as uncontrolled diabetes, uncontrolled hypertension, active clinically serious infection > CTCAE Grade 2, history of bleeding diathesis or coagulopathy, impairment of GI function or GI disease that may significantly alter absorption of the study regimen (i.e. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow tablets).
* Thrombolic or embolic events such as cerebrovascular accident including transient ischemic attacks within past 6 months
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of 1st dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of 1st dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of 1st study drug.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Pt is < 3 years free of another primary malignancy except: if other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is basal cell skin cancer or cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Pts unwilling or unable to comply with protocol including ability to swallow whole pills or presence of any malabsorption syndrome.
* Concurrent administration of St. John's Wort.
* Clinically serious infection requiring active intervention (CTCAE grade 2 or greater).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Result] Reardon DA, Vredenburgh JJ, Desjardins A, Peters K, Gururangan S, Sampson JH, Marcello J, Herndon JE 2nd, McLendon RE, Janney D, Friedman AH, Bigner DD, Friedman HS. Effect of CYP3A-inducing anti-epileptics on sorafenib exposure: results of a phase II study of sorafenib plus daily temozolomide in adults with recurrent glioblastoma. J Neurooncol. 2011 Jan;101(1):57-66. doi: 10.1007/s11060-010-0217-6. Epub 2010 May 5. PMID 20443129

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib + Temozolomide: Subjects receive 400mg of Sorafenib twice daily and 50mg/m^2 of Temozolomide once daily
  Subjects continue to receive treatment until any of the following: progressive disease, unacceptable toxicity, non-compliance with study guidelines, withdrawal of patient consent, intercurrent non-cancer-related illness that prevents continuation of therapy or regular follow-up, general or specific changs in a subject's condition which render the patient unacceptable for treatment in the judgement of the investigator, or study closure
Period: Overall Study
Arm/Group | Sorafenib + Temozolomide
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib + Temozolomide
Number analyzed (Participants) | 32
Age Continuous [Median (Full Range); unit: years] | 53.6 [30.4 to 72.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression Free Survival (PFS)
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Macdonald criteria, or to death due to any cause.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Sorafenib + Temozolomide
Number analyzed (Participants) | 32
percentage of patients | 9.4 [2.4 to 22.3]

2. Secondary Outcome: Safety and Toxicity of Combination
Description: Number of participants experiencing a toxicity of at least grade 3 that was deemed possibly, probably, or definitely related to the treatment.
Time Frame: 16 months
Measure: Number; unit: participants
Arm/Group | Sorafenib + Temozolomide
Number analyzed (Participants) | 32
participants | 19

3. Secondary Outcome: Pharmacokinetics: C-max
Description: Blood sampling for sorafenib pharmacokinetics was performed on days 1 and 28 of cycle 1 and was obtained before and at 0.5, 1, 2, 4, 6, 8, and 24 h after the morning dose. C-max refers to maximum plasma concentration. The pharmacokinetics of those patients taking enzyme-inducing antiepileptic drugs (EIAED) and those who were not were analyzed separately.
Time Frame: 13 months
Population: 9 participants who were on EIAEDs had 24 hour sorafenib concentration versus time profiles from both day 1 and day 28 of cycle 1. 14 participants who were not on EIAEDs underwent similar assessment for day 1 but only 10 of these participants had samples available for day 28 measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/L
Groups:
- EIAEDs-Day 1: Blood samples taken on day 1 of cycle 1 from patients currently taking EIAEDs.
- EIAEDs-Day 28: Blood samples taken on day 28 of cycle 1 from patients currently taking EIAEDs.
- Non-EIAEDs-Day 1: Blood samples taken on day 1 of cycle 1 from patients not currently taking EIAEDs.
- Non-EIAEDs-Day 28: Blood samples taken on day 28 of cycle 1 from patients not currently taking EIAEDs.
Arm/Group | EIAEDs-Day 1 | EIAEDs-Day 28 | Non-EIAEDs-Day 1 | Non-EIAEDs-Day 28
Number analyzed (Participants) | 9 | 9 | 14 | 10
ug/L | 3397.3 (66.8) | 3813.9 (40.7) | 3155.1 (41.7) | 8118.8 (60.8)

4. Secondary Outcome: Pharmacokinetics: T-max
Description: Blood sampling for sorafenib pharmacokinetics was performed on days 1 and 28 of cycle 1 and was obtained before and at 0.5, 1, 2, 4, 6, 8, and 24 h after the morning dose. T-max refers to time to maximum concentration. The pharmacokinetics of those patients taking enzyme-inducing antiepileptic drugs (EIAED) and those who were not were analyzed separately.
Time Frame: 13 months
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | EIAEDs-Day 1 | EIAEDs-Day 28 | Non-EIAEDs-Day 1 | Non-EIAEDs-Day 28
Number analyzed (Participants) | 9 | 9 | 14 | 10
hours | 8.2 [2.0 to 24.7] | 2.1 [0 to 2.3] | 24.0 [2.0 to 25.5] | 4.2 [0 to 8.2]

5. Secondary Outcome: Pharmacokinetics: AUC-24
Description: Blood sampling for sorafenib pharmacokinetics was performed on days 1 and 28 of cycle 1 and was obtained before and at 0.5, 1, 2, 4, 6, 8, and 24 h after the morning dose. AUC-24 refers to area under the plasma concentration-time curve from 0 to 24 hours. The pharmacokinetics of those patients taking enzyme-inducing antiepileptic drugs (EIAEDs) and those who were not were analyzed separately.
Time Frame: 13 months
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*H/L
Arm/Group | EIAEDs-Day 1 | EIAEDs-Day 28 | Non-EIAEDs-Day 1 | Non-EIAEDs-Day 28
Number analyzed (Participants) | 9 | 9 | 14 | 10
ug*H/L | 45309.7 (61.8) | 47148.2 (65.7) | 45238.7 (44.1) | 128820.8 (73.2)

ADVERSE EVENTS:
Time Frame: 16 months
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov
Arm/Group | Sorafenib + Temozolomide
Serious Adverse Events (participants affected / at risk) | 4/32
Other Adverse Events (participants affected / at risk) | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Temozolomide (N=32)
Pancreatitis (Gastrointestinal disorders) | 2
Lung infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lipase increased (Investigations) | 2
Serum amylase increased (Investigations) | 2
Seizure (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Temozolomide (N=32)
Anemia (Blood and lymphatic system disorders) | 2
Blurred vision (Eye disorders) | 5
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 7
Lung infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Lipase increased (Investigations) | 8
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 3
Serum amylase increased (Investigations) | 2
White blood cell decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Ataxia (Nervous system disorders) | 5
Cognitive disturbance (Nervous system disorders) | 6
Depressed level of consciousness (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysphasia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 6
Peripheral motor neuropathy (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Reproductive system and breast disorders - Other, specify: Sexual Dysfunction (Reproductive system and breast disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No